CLINICAL TRIAL: NCT05233397
Title: Phase 2 Study of Systemic IL-6 Receptor Antagonist ACTEMRA® (Tocilizumab) for the Treatment of Progressive/Recurrent Pediatric Adamantinomatous Craniopharyngioma
Brief Title: ACTEMRA® for the Treatment of Pediatric Adamantinomatous Craniopharyngioma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CONNECT1905
Record Dates: First submitted 2022-01-25; First posted 2022-02-10 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-02

CONDITIONS: Adamantinomatous Craniopharyngioma; Recurrent Adamantinomatous Craniopharyngioma
MeSH Terms: conditions — Craniopharyngioma | interventions — tocilizumab

STUDY DESIGN:
Intervention Model Description: ACTEMRA® (tocilizumab)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Stratum 1 and Stratum 2 (Experimental): Stratum 1: Patients with progressive or recurrent adamantinomatous craniopharyngiomas following radiation therapy.
  Stratum 2: Patients with measurable adamantinomatous craniopharyngioma who have undergone surgery but have not previously received radiation therapy. Progressive disease is allowed but not required
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — For < 30 kg: 12 mg/kg IV every 2 weeks; For ≥30 kg: 8 mg/kg IV every 2 weeks
  Other Names: ACTEMRA®

SUMMARY:
ACTEMRA (tocilizumab) is an IL-6 receptor antagonist used for the treatment of adult Rheumatoid Arthritis as well as Polyarticular (PJIA) and Systemic (SJIA) Juvenile Idiopathic Arthritis. In this Phase II, the drug will be used to treat pediatric patients diagnosed with recurrent Adamantinomatous Craniopharyngioma including patients who have undergone surgery and/or radiation therapy.

DETAILED DESCRIPTION:
Adamantinomatous Craniopharyngioma (ACP) is a highly debilitating pediatric brain tumor that lacks medical anti-tumor therapies. Current therapy, which depends largely on surgery and radiation, is associated with poor quality of life and becomes more challenging and risky in the setting of recurrent disease. Recent discoveries regarding the biological characteristics of ACP indicate that available agents, including IL-6 pathway blockers may have efficacy in the control of ACP. We hypothesize that the IL6- receptor antagonist ACTEMRA (tocilizumab) will be safe and effective at inducing tumor response in children with residual ACP.

In this study, up to 38 patients will receive tocilizumab at the dose approved for pediatric Systemic Juvenile Idiopathic Arthritis (< 30 kg: 12 mg/kg IV every 2 weeks; ≥30 kg: 8 mg/kg IV every 2 weeks). Therapy may continue for up to two years (26 cycles).

It will be a multi-center Phase 2 trial with two strata for patients aged >1 year and <25 years with unresectable ACP who may have been previously treated with radiation (Stratum 1, 18 patients) or without radiation (Stratum 2, 18 patients).

ELIGIBILITY:
Inclusion Criteria:

1. Age: Patients must be ≥ 12 months and ≤ 39 years of age at the time of study enrollment.
2. Diagnosis: Patients with histologically-confirmed adamantinomatous craniopharyngioma (ACP) Histologic confirmation of ACP may be made on solid tumor or, if no solid tumor can be safely obtained, cyst fluid with classic ACP characteristics of thick, cholesterol-rich, greenish-brown liquid in the context of imaging features consistent with craniopharyngioma, including lobulated, cystic/solid mass with calcifications that originates in the sellar/suprasellar region.
3. Disease Status: Patients must have measurable disease.

   * Stratum 1: Patients with progressive or recurrent ACP who demonstrate cystic and/or solid recurrence or progression at least 6 months post completion of radiation therapy
   * Stratum 2: Patients with measurable ACP who have undergone surgery but have NOT previously undergone irradiation (but may have received prior systemic or intracystic therapy). Progressive disease is allowed but not required.
4. Performance Level: Karnofsky ≥ 50% for patients > 16 years of age and Lansky ≥ 50 for patients ≤ 16 years of age (See Appendix I). Note: Neurologic deficits in patients with CNS tumors must have been stable for at least 7 days prior to study enrollment. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
5. Prior Therapy: Patients must have recovered or stabilized from the acute toxic effects of prior treatments

   * Biologic (anti-neoplastic agent): At least 7 days must have elapsed after the last (systemic or intracystic) dose of a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair
   * Immunotherapy: At least 42 days after the completion of any type of systemic immunotherapy, e.g. tumor vaccines.
   * Monoclonal antibodies: At least 21 days after the last dose of a monoclonal antibody.
   * Radiation therapy: Patients must have had their last (conventional or hypofractionated) fraction of: a) Focal irradiation > 6 months prior to enrollment and b) No prior craniospinal irradiation is permitted.
   * Corticosteroids: Patients receiving dexamethasone must be on a stable or decreasing dose for at least 1 week prior to enrollment
   * Myelosuppressive systemic therapy: At least 21 days must have elapsed after the last systemic myelosuppressive therapy.
   * Surgery: At least 6 weeks must have elapsed since major or intermediate surgery. Major surgery includes major craniotomy for tumor resection or cyst fenestration, organ resection, exploratory laparotomy. Intermediate procedures include ventriculoperitoneal shunt placement, stereotactic brain biopsy and intraventricular catheter placement. Minor procedures that are not excluded include skin biopsy/incision and drainage, bone marrow aspirate, and central venous catheter placement. Ommaya aspirations and Lumbar Punctures are considered minor procedures..
6. Organ Function Requirements

   Adequate Bone Marrow Function Defined as:
   * Peripheral absolute neutrophil count (ANC) ≥1000/mm3
   * Platelet count ≥100,000/mm3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
   * Hemoglobin >8 g/dL (may be transfused)

   Adequate Renal Function Defined as:
   * Creatinine clearance or radioisotope GFR > 70ml/min/1.73 m2 or
   * A serum creatinine based on (Schwartz et al. J. Peds, 106:522, 1985) age/gender as follows:

     1 to < 2 years: maximum serum creatinine 0.6 mg/dL for males and females. 2 to < 6 years: maximum serum creatinine 0.8 mg/dL for males and females. 6 to < 10 years: maximum serum creatinine 1.0 mg/dL for males and females. 10 to < 13 years: maximum serum creatinine 1.2 mg/dL for males and females. 13 to < 16 years: maximum serum creatinine 1.5 mg/dL for males and 1.4 mg/dL for females.

     ≥ 16 years: maximum serum creatinine 1.7 mg/dL for males and 1.4 mg/dL for females.

   Adequate Liver Function Defined as:
   * Total bilirubin within normal institutional limits
   * AST (SGOT) ≤ 2.5 × institutional upper limit of normal
   * ALT (SGPT) ≤ 2.5 × institutional upper limit of normal

   Adequate Neurologic Function Defined as:
   * Patients with neurological deficits should have deficits that are stable for a minimum of 1 week prior to enrollment.
   * Patients with current seizure disorders may be enrolled if seizures are well-controlled on antiepileptic therapies.
7. Informed Consent: All patients and/or their parents or legally authorized representatives must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.

Exclusion Criteria:

1. Pregnancy or Breast-Feeding: Pregnant or breast-feeding women will not be entered on this study due to unknown risks of fetal and teratogenic adverse events as seen in animal/human studies. Pregnancy tests must be obtained in girls who are post-menarchal. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method for at least 90 days after discontinuation of drug for females and at least 60 days for males. For females of childbearing potential, agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods (bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices; hormonal contraceptive methods must be supplemented by a barrier method) and agreement to refrain from donating eggs are required. For males of reproductive potential, agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm.
2. Gastrointestinal Disease: Patients with a history of serious gastrointestinal disease, including inflammatory bowel disease or gastrointestinal perforation
3. Concomitant Medications

   * Corticosteroids: Patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are not eligible.
   * Investigational Drugs: Patients who are currently receiving another investigational drug are not eligible.
   * Anti-cancer Agents: Patients who are currently receiving other anti-cancer agents are not eligible.
4. Study Specific:

   * Patients who have an uncontrolled infection are not eligible.
   * Patients who have received any live or attenuated vaccinations within three months prior to start of therapy are not eligible.
   * Any significant concurrent medical or surgical condition that would jeopardize the patient's safety or ability to complete the study, including, but not limited to, disease of the nervous, renal, hepatic, cardiac (such as symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia), pulmonary, or endocrine system
   * Patients who have a history of Human Immunodeficiency Virus, Hepatitis B Virus, Hepatitis C Virus or Tuberculosis infection are not eligible.
   * Patients who have received a prior solid organ transplantation are not eligible.
   * Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible.
   * Patients who have a history of alcohol, drug, or chemical abuse within 6 months of screening.
   * Patients who have had major or intermediate surgery within the last 6 weeks or who have concerns for poor postsurgical wound healing.
   * Patients who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to tocilizumab and its excipients are not eligible.

Ages: 1 Year to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-12-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Sustained objective response rate of patients with recurrent/progressive previously irradiated ACP to treatment with systemic tocilizumab | From Day 1 of treatment through 30 days following end of protocol treatment
  To calculate the number of patients who experience sustained objective response rate [minor response (MR) + partial response (PR) + complete response (CR)] of patients with recurrent/progressive previously irradiated Adamantinomatous Craniopharyngioma to treatment with systemic tocilizumab (Stratum 1).
Sustained objective response rate of patients with measurable ACP who have undergone surgery but have not been previously treated with radiation to treatment with systemic tocilizumab | From Day 1 of treatment through 30 days following end of protocol treatment
  To calculate the number of patients who experience sustained objective response rate (MR + PR + CR) of patients with measurable Adamantinomatous Craniopharyngioma who have undergone surgery but have not been previously treated with radiation to treatment with systemic tocilizumab (Stratum 2).

SECONDARY OUTCOMES:
Biological effects of tocilizumab on ACP tumor tissue and cyst fluid. | From Day 1 of treatment through 30 days following end of protocol treatment
  To measure the concentrations of IL-6, IL-8, IL-10, CXCL1, CXCR2, IDO-1 and IL-6R using a combination of ELISA, RNAseq, immunohistochemistry and immunofluorescence in cyst fluid or tumor tissue or blood. Comparisons will be made with known levels in the literature and among patient samples from within the study.
Toxicities associated with tocilizumab in children with ACP | From Day 1 of treatment through 30 days following end of protocol treatment
  To calculate the number of participants with, as well as frequency and severity of, tocilizumab-related Adverse Events as assessed by CTCAE v5.0 in children with recurrent or refractory ACP.
PFS of ACP patients treated with tocilizumab after radiation | 12 months
  To assess one-year progression-free survival (PFS) rates for patients with ACP who are treated with tocilizumab following progression after radiation (Stratum 1).
PFS of ACP patients treated with tocilizumab who have not received radiation | 12 months
  To assess one-year progression-free survival (PFS) rates for patients with ACP who are treated with tocilizumab who have not previously received radiation (Stratum 2).

CONTACTS AND LOCATIONS:
Overall Officials: Holly Lindsay, MD, Study Chair — Children's Hospital Colorado; Todd C Hankinson, MD, Study Chair — Children's Hospital Colorado; Maryam Fouladi, MD, Principal Investigator — Nationwide Children's Hospital
Locations (12):
- United States (8):
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Nicklaus Children's Hospital, Miami, Florida
  - Duke Children's Hospital, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Australia (3):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Perth Children's Hospital, Perth, Western Australia
- McGill University Health Center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Editorial: Iron and folate deficiency in pregnancy. Med J Aust. 1974 Sep 28;2(13):470-1. No abstract available. PMID 4431348
- [Background] Gottschalk ME, Kemp RG. Interaction of dinucleotides with muscle phosphofructokinase. Biochemistry. 1981 Apr 14;20(8):2245-51. doi: 10.1021/bi00511a027. No abstract available. PMID 6263310
- [Background] Choy EH, Isenberg DA, Garrood T, Farrow S, Ioannou Y, Bird H, Cheung N, Williams B, Hazleman B, Price R, Yoshizaki K, Nishimoto N, Kishimoto T, Panayi GS. Therapeutic benefit of blocking interleukin-6 activity with an anti-interleukin-6 receptor monoclonal antibody in rheumatoid arthritis: a randomized, double-blind, placebo-controlled, dose-escalation trial. Arthritis Rheum. 2002 Dec;46(12):3143-50. doi: 10.1002/art.10623. PMID 12483717
- [Background] De Benedetti F, Brunner HI, Ruperto N, Kenwright A, Wright S, Calvo I, Cuttica R, Ravelli A, Schneider R, Woo P, Wouters C, Xavier R, Zemel L, Baildam E, Burgos-Vargas R, Dolezalova P, Garay SM, Merino R, Joos R, Grom A, Wulffraat N, Zuber Z, Zulian F, Lovell D, Martini A; PRINTO; PRCSG. Randomized trial of tocilizumab in systemic juvenile idiopathic arthritis. N Engl J Med. 2012 Dec 20;367(25):2385-95. doi: 10.1056/NEJMoa1112802. PMID 23252525
- [Background] Donson AM, Apps J, Griesinger AM, Amani V, Witt DA, Anderson RCE, Niazi TN, Grant G, Souweidane M, Johnston JM, Jackson EM, Kleinschmidt-DeMasters BK, Handler MH, Tan AC, Gore L, Virasami A, Gonzalez-Meljem JM, Jacques TS, Martinez-Barbera JP, Foreman NK, Hankinson TC; Advancing Treatment for Pediatric Craniopharyngioma Consortium. Molecular Analyses Reveal Inflammatory Mediators in the Solid Component and Cyst Fluid of Human Adamantinomatous Craniopharyngioma. J Neuropathol Exp Neurol. 2017 Sep 1;76(9):779-788. doi: 10.1093/jnen/nlx061. PMID 28859336
- [Background] Fischer E, Varga F. Effect of taurocholate pretreatment on the biliary excretion of exogenous organic anions in rats. Arch Int Pharmacodyn Ther. 1984 Feb;267(2):187-99. PMID 6712354
- [Background] Storozhuk VM. [Functional properties of neurons of the somato-sensory cortex, activated by stimulation of the pyramidal tract]. Zh Vyssh Nerv Deiat Im I P Pavlova. 1968 Jul-Aug;18(4):681-90. No abstract available. Russian. PMID 5718945
- [Background] Mihara M, Kasutani K, Okazaki M, Nakamura A, Kawai S, Sugimoto M, Matsumoto Y, Ohsugi Y. Tocilizumab inhibits signal transduction mediated by both mIL-6R and sIL-6R, but not by the receptors of other members of IL-6 cytokine family. Int Immunopharmacol. 2005 Nov;5(12):1731-40. doi: 10.1016/j.intimp.2005.05.010. PMID 16102523
- [Background] Wood MJ, Hennigan DB. Radionuclide tagged red blood cells in the gallbladder. Clin Nucl Med. 1984 May;9(5):289-90. doi: 10.1097/00003072-198405000-00013. No abstract available. PMID 6086204
- [Background] Nishimoto N, Kishimoto T. Inhibition of IL-6 for the treatment of inflammatory diseases. Curr Opin Pharmacol. 2004 Aug;4(4):386-91. doi: 10.1016/j.coph.2004.03.005. PMID 15251133
- [Background] Nishimoto N, Kishimoto T. Humanized antihuman IL-6 receptor antibody, tocilizumab. Handb Exp Pharmacol. 2008;(181):151-60. doi: 10.1007/978-3-540-73259-4_7. PMID 18071945
- [Background] Nishimoto N, Yoshizaki K, Maeda K, Kuritani T, Deguchi H, Sato B, Imai N, Suemura M, Kakehi T, Takagi N, Kishimoto T. Toxicity, pharmacokinetics, and dose-finding study of repetitive treatment with the humanized anti-interleukin 6 receptor antibody MRA in rheumatoid arthritis. Phase I/II clinical study. J Rheumatol. 2003 Jul;30(7):1426-35. PMID 12858437
- [Background] Nishimoto N, Yoshizaki K, Miyasaka N, Yamamoto K, Kawai S, Takeuchi T, Hashimoto J, Azuma J, Kishimoto T. Treatment of rheumatoid arthritis with humanized anti-interleukin-6 receptor antibody: a multicenter, double-blind, placebo-controlled trial. Arthritis Rheum. 2004 Jun;50(6):1761-9. doi: 10.1002/art.20303. PMID 15188351
- [Background] Sato K, Tsuchiya M, Saldanha J, Koishihara Y, Ohsugi Y, Kishimoto T, Bendig MM. Reshaping a human antibody to inhibit the interleukin 6-dependent tumor cell growth. Cancer Res. 1993 Feb 15;53(4):851-6. PMID 8428365
- [Background] Yokota S, Miyamae T, Imagawa T, Iwata N, Katakura S, Mori M, Woo P, Nishimoto N, Yoshizaki K, Kishimoto T. Therapeutic efficacy of humanized recombinant anti-interleukin-6 receptor antibody in children with systemic-onset juvenile idiopathic arthritis. Arthritis Rheum. 2005 Mar;52(3):818-25. doi: 10.1002/art.20944. PMID 15751095